CLINICAL TRIAL: NCT02730026
Title: Comparison of the Clinical Efficacy of Ketoprofen, Associated or Not With Omeprazole, in the Control of Pain, Swelling and Trismus in Lower Third Molar Removal
Brief Title: Comparison of the Clinical Efficacy of Ketoprofen, Associated or Not With Omeprazole in Lower Third Molar Removal
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Luis Fernando Simoneti (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor-Investigator, Luis Fernando Simoneti, DDS, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 44808215.6.0000.5417
Record Dates: First submitted 2015-09-10; First posted 2016-04-06 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Pain; Other Surgical Procedures
Keywords: Ketofrofen; Omeprazole; Lower Third Molar; Oral Surgery
MeSH Terms: conditions — Pain | interventions — Ketoprofen; Omeprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Surgery with Ketoprofen (Experimental): Fifty healthy volunteers underwent removal one of lower third molar, will be treated to control pain, swelling and trismus with ketoprofen 100 mg
  Interventions: Drug: Ketoprofen
- Surgery with Ketoprofen and Omeprazole (Experimental): Fifty healthy volunteers underwent removal the other lower third molars, will be treated to control pain, swelling and trismus with ketoprofen 200 mg associated with Omeprazole 20 mg
  Interventions: Drug: Ketoprofen and Omeprazole

INTERVENTIONS:
Drug: Ketoprofen — Clinical efficacy of the Ketoprofen 100 mg was study after lower third molar surgery.
  Other Names: Lower third molar surgery with Ketoprofen
  Arms: Surgery with Ketoprofen
Drug: Ketoprofen and Omeprazole — Clinical efficacy of the Ketoprofen 200 mg and Omeprazole 20 mg will be study after lower third molar surgery.
  Other Names: Lower third molar surgery with Ketoprofen and Omeprazole
  Arms: Surgery with Ketoprofen and Omeprazole

SUMMARY:
The control of pain, swelling and trismus in patients undergoing oral and maxillofacial surgery is frequently performed through the administration of non-steroidal anti-inflammatory drugs (NSAIDS). The present study aims to evaluate in a double blind, randomized and crossover manner the clinical efficacy of ketoprofen (immediate release - 100 mg) and ketoprofen in association with omeprazole (modified release - 200 mg ketoprofen with 20 mg omeprazole) in 50 patients aged 18 years or older that require removal of both lower third molars symmetrically positioned. After collection, data will be analyzed by means of graphs and tables to allow the appropriate analyses. Paired t-test will be used to compare the duration of surgeries. Nonparametric Wilcoxon test will be used for the analysis of "rescue medication" and postoperative pain parameters (visual analog scale). Data of "mouth opening" and "swelling" will be statistically analyzed through analysis of variance (ANOVA) followed by Tukey's test for multiple comparisons. Statistical significance will be set at 5%. Results will be presented as mean ± standard deviation of the mean.

DETAILED DESCRIPTION:
Studies have shown that NSAIDS exert their therapeutic effect by the inhibition of cyclooxigenases (COX) 1 and 2, which determines the inhibition of prostaglandins production whose effects potentiate the action of many inflammatory mediators. The protocol for the administration of these formulations will involve the administration of a tablet of the immediate release product (100 mg) every 12 hours, and one capsule of the modified release product (200 mg ketoprofen with omeprazole) every 24 hours, during 4 days.

The following parameters will be analyzed:

1. subjective postoperative pain evaluation, with the aid of a visual analogue scale,
2. mouth opening before the surgery, on the 2nd and 7th postoperative days (moment of suture removal),
3. beginning and duration of the surgery after anesthetic administration,
4. incidence, type and severity of adverse reactions,
5. total amount of rescue analgesic medication (paracetamol),
6. facial swelling measured on the 2nd and 7th postoperative days (in comparison with the measurements before the surgery).

ELIGIBILITY:
Inclusion Criteria:

* Need of lower third molar surgeries in similar positions

Exclusion Criteria:

* Presence of systemic diseases;
* Presence of local inflammation and/or infection;
* Any history of allergic reaction to local anesthetics, gastrointestinal bleeding or ulceration;
* Cardiovascular, kidney or hepatic diseases;
* Patients who are making use of antidepressants, diuretics or anticoagulants;
* Asthma and allergy to aspirin, naproxen or any other nonsteroidal antiinflammatory drug;
* Regular use of any nonsteroidal antiinflammatory drug, pregnancy or breast feeding.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Subjective evaluation of postsurgical pain | Fourth postoperative hour
  Subjective evaluation of postsurgical pain, which was annotated by the volunteer, a Visual Analogue Scale (VAS, 0-100 mm) at the fourth postoperative hour.
Quality of anesthesia during surgery based on a category 3point scale | During the surgical procedure
  Quality of anesthesia during surgery based on a category 3point scale: 1) the patient reported no discomfort; 2) the patient reported discomfort, without the need to supplement the anesthesia; 3) reported some discomfort by the patient, requiring anesthesia complementation. Intraoral bleeding that will be evaluated by the surgeon according to a 3point scale (1: minimal, 2: normal and 3: Maximum), immediately after the following steps: injection of the first cartridge anesthesia, incision, mucoperiosteal detachment, osteotomies, tooth section, extraction, cleaning and suturing.
Intraoperative bleeding, rated by the surgeon according to a 3 point category rating scale | During the surgical procedure
  Intraoperative bleeding, rated by the surgeon according to a 3 point category rating scale (1 minimal bleeding; 2 normal bleeding; 3 excessive bleeding) (SISK, 1986), immediately after the following steps: injection of the first cartridge of articaine, tissue incision, flap reflection, bone removal (when this procedure was necessary), tooth extraction, cleaning of the operated site, and completion of suturing.
Heart rate | During the surgical procedure
  Median heart rate to be verified and recorded surgical at moments described above, carried out with the aid of a system for monitoring hemodynamic parameters
Oxygen saturation | During the surgical procedure
  Median oxygen saturation recorded at surgical moments described above, carried out with the aid of a system for monitoring hemodynamic parameters.
Systolic blood pressure | During the surgical procedure
  Median systolic blood pressure to be verified and recorded at surgical moments previously described (injection of the first cartridge anesthesia, incision, mucoperiosteal detachment, osteotomies, tooth section, extraction, cleaning and suturing), carried out with the aid of a system for monitoring hemodynamic parameters
Diastolic blood pressure | During the surgical procedure
  Median diastolic blood pressure to be verified and recorded at surgical moments previously described (injection of the first cartridge anesthesia, incision, mucoperiosteal detachment, osteotomies, tooth section, extraction, cleaning and suturing), carried out with the aid of a system for monitoring hemodynamic parameters

SECONDARY OUTCOMES:
Mouth opening (mm) between the mesial-incisal corners of the upper and lower right central incisors at maximum opening of the jaws | Second and Seventh postoperative days
  Mouth opening (mm) between the mesial-incisal corners of the upper and lower right central incisors at maximum opening of the jaws was measured and recorded before the surgery and during the second and seventh postoperative days.
Onset and duration of surgery after administration of anesthetic | During the surgery
  Will only be considered those surgeries in which there is no long time gap between the two surgical times.
Incidence, type and severity of adverse reactions | Seventh postoperative day
  Will be considered as adverse reactions: gastrointestinal irritation, nausea, vomiting, bleeding, allergy, headache, dizziness, drowsiness or any other type of reaction presented after surgery.
Total amount of rescue medication | Seventh postoperative day
  The total amount of rescue medication that was used by the patient during the postoperative period (paracetamol 750 mg) will be analyzed
Measurement the facial edema distance between the lateral corner of the eye and the gonion, away from the tragus corner of the mouth and away from the tragus to the soft tissue of pogonion. | On the second day after surgery and on the seventh day after surgery
  It will apply the method used by Ustun et al. (2003), which takes into account the sum of the following measures (obtained with flexible tape measure): A) distance between the lateral corner of the eye and the gonion, B) away from the tragus corner of the mouth and C) away from the tragus to the soft tissue of pogonion. Preoperative sum of three measures will be considered as the baseline that way. The difference between the values obtained in the postoperative period and baseline indicate the facial edema in the 2nd and 7th days.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Fernando Simoneti, DDS, Principal Investigator — University of Sao Paulo
Locations (1):
- University of Sao Paulo, Bauru, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided